CLINICAL TRIAL: NCT00358670
Title: A Long-Term Efficacy and Safety Study of Infliximab in the Treatment of Moderate to Severe Plaque-Type Psoriasis
Brief Title: Long-Term Effects of Infliximab in the Treatment of Moderate to Severe Psoriasis [Extension of Study P04271, NCT00251641] (P04563)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Infusion reactions during re-induction cycles after a period of no treatment. Please see "Purpose" section.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04563; EUDRACT NUMBER:2005-005367-28
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance Infliximab (Active Comparator): Infliximab 5 mg/kg by body weight every 8 weeks
  Interventions: Biological: infliximab
- Intermittent Infliximab (Experimental): Infliximab 5 mg/kg by body weight at Weeks 0, 2, 6 and 14 following a 50% reduction in Psoriasis Area and Severity Index (PASI) from the Study P04271 Baseline
  Interventions: Biological: infliximab

INTERVENTIONS:
Biological: infliximab — Infliximab maintenance therapy
  intravenous (IV) infusion every 8 weeks, 5 mg/kg body weight (first infusion at Week 4/Visit 2).
  Other Names: SCH 215596; Remicade
  Arms: Maintenance Infliximab
Biological: infliximab — Infliximab intermittent therapy:
  Paricipants will receive no infliximab treatment until the Week 26 improvement in PASI from Baseline (original Study P04271 [NCT00251641] Baseline) is reduced by more than 50%. At that time, participants will receive an infliximab infusion, 5 mg/kg body weight. Participants may receive additional infusions at 0, 2, 6, and 14 weeks after the first infusion of the cycle (ie, a maximum of 4 infusions in each infusion cycle) as needed until they respond, defined as a >=75% improvement in PASI from the original Baseline in Study P04271. Subjects will receive no further treatment until they relapse again (ie, improvement in PASI from Baseline is reduced by more than 50%), at which time participants will receive another infusion cycle of up to 4 infusions, as described above. Throughout the study, intermittent treatment infusion cycles will be repeated whenever participants relapse.
  Other Names: SCH 215596; Remicade
  Arms: Intermittent Infliximab

SUMMARY:
This is a long-term, randomized, multi-center, open-label study of infliximab treatment in adults with moderate to severe plaque-type psoriasis. This study is the long-term extension of Study P04271 (NCT00251641); Study P04271 is a Phase 3b, randomized, parallel-group, multicenter, open-label, 26-week study comparing the efficacy and safety of infliximab versus methotrexate in the treatment of adult subjects with moderate to severe plaque-type psoriasis. The objectives of this study are to assess the efficacy and safety of long-term maintenance therapy versus intermittent therapy with 5 mg/kg infliximab in a moderate to severe plaque-type psoriasis population.

During an interim safety evaluation of the trial, a higher incidence of serious and severe infusion reactions was observed in the intermittent treatment arm, consisting of a re-induction cycle (maximum of 4 infusions at 0, 2, 6 and 14 weeks) after a period of no treatment compared with the maintenance arm (infusions every 8 weeks without an interruption of treatment). Consequently, the sponsor has terminated the trial. The label will be updated to reflect this new information relating to the use of a re-induction regimen with infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have met all inclusion/exclusion criteria in Study P04271 (NCT00251641).
* Subjects must have been originally randomized to infliximab in Study P04271.
* Subjects must have completed the full 26 weeks of Study P04271.
* Subjects must have remained on infliximab for the full 22 weeks of treatment in Study P04271.
* Subjects must have achieved an improvement in Psoriasis Area and Severity Index (PASI) score >=75% from Baseline of Study P04271 to Week 26 of Study P04271.
* Subjects must agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study.
* Subjects are considered eligible according to the following tuberculosis (TB) criteria:

  * Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination;
  * Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study medication.
* Subjects' Baseline (Visit 1) clinical laboratory tests (complete blood count, blood chemistry, and urinalysis) must be within the following parameters:

  * Hemoglobin >=10 g/dL
  * White blood cells >=3.5 x 10^9/L
  * Neutrophils >=1.5 x 10^9/L
  * Platelets >=100 x 10^9/L
  * Serum creatinine <1.5 mg/dL (or <133 umol/L)
  * Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, and gamma-glutamyltransferase levels as outlined in Protocol P04563.
  * Total bilirubin <2 x upper limit of normal [Note: If Baseline laboratory tests are not yet available, then the previous laboratory tests from Week 22 of the parent study (Study P04271) should be used for enrollment. When the Baseline laboratory tests become available, the investigator must apply the above parameters to determine a subject's eligibility.]
* Subjects must be free of any clinically significant disease (other than plaque-type psoriasis or psoriatic arthritis) that would interfere with the study evaluations.
* Subjects must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Women of childbearing potential and all men must be using adequate birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) and must continue using such measures until 6 months after receiving the last infusion of study medication.
* Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline.

Exclusion Criteria:

* Subjects who have any significant ongoing adverse events (AEs) or AEs from Study P04271 (NCT00251641) that would prohibit further treatment with infliximab at the time of entry.
* Subjects originally randomized to methotrexate or subjects who received methotrexate at any time during their participation in Study P04271.
* Subjects who have non-plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular).
* Subjects who have current drug-induced psoriasis (eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Female subjects who are pregnant, nursing, and both men and women who are planning pregnancy during the study period or during the 6 months after receiving of the last infusion of study medication.
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subjects who are staff personnel directly involved with this study.
* Subjects who are family members of the investigational study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Reich K, Wozel G, Zheng H, van Hoogstraten HJ, Flint L, Barker J. Efficacy and safety of infliximab as continuous or intermittent therapy in patients with moderate-to-severe plaque psoriasis: results of a randomized, long-term extension trial (RESTORE2). Br J Dermatol. 2013 Jun;168(6):1325-34. doi: 10.1111/bjd.12404. PMID 23621698

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent Infliximab: Infliximab 5 mg/kg by body weight at Weeks 0, 2, 6 and 14 following a 50% reduction in Psoriasis Area and Severity Index (PASI) from the Study P04271 (NCT00251641) Baseline
Period: Overall Study
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Started | 222 | 219
Completed | 0 | 0
Not Completed | 222 | 219
Not completed — Adverse Event | 26 | 29
Not completed — Lack of Efficacy | 20 | 23
Not completed — Protocol Violation | 6 | 9
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 13 | 24
Not completed — Protocol Defined Clinical Event | 0 | 1
Not completed — Did Not Meet Protocol Eligibility | 0 | 3
Not completed — Administrative | 153 | 125

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Infliximab: Infliximab 5 mg/kg by body weight at Weeks 0, 2, 6 and 14 following a 50% reduction in PASI from the Study P04271 (NCT00251641) Baseline
- Total: Total of all reporting groups
Arm/Group | Maintenance Infliximab | Intermittent Infliximab | Total
Number analyzed (Participants) | 222 | 219 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.1) | 43.3 (12.2) | 44.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 63 | 133
  Male | 152 | 156 | 308

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Psoriasis Area and Severity Index 75 (PASI75) Response at Week 128
Description: PASI75 defined as the number of participants who achieved a >=75% improvement in Psoriasis Area and Severity Index (PASI) from the original Baseline in Study P04271 (NCT00251641).
Time Frame: 128 weeks
Population: Due to the early termination of the study, no subjects completed 128 weeks of therapy.
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Who Achieved PASI75 Response at Week 52
Description: PASI75 defined as the number of participants who achieved a >=75% improvement in PASI from the original Baseline in Study P04271 (NCT00251641)
Time Frame: 52 weeks
Population: Descriptive summary of all randomized subjects who completed 52 weeks (+ or - 4 weeks) of therapy. Based on best (minimum) PASI score at Week 52.
Measure: Number; unit: Participants
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Number analyzed (Participants) | 101 | 83
Participants | 81 | 39

3. Secondary Outcome: Number of Participants Who Achieved PASI75 Response at Week 100
Description: as for outcome 2
Time Frame: 100 Weeks
Population: Descriptive summary of all randomized subjects who completed 100 weeks (+ or - 4 weeks) of therapy. Based on best (minimum) PASI score at Week 100.
Measure: Number; unit: Participants
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Number analyzed (Participants) | 21 | 13
Participants | 18 | 9

4. Secondary Outcome: PASI 6-month Area Under the Curve (AUC); (Time Adjusted Total PASI Score Over the 6 Month Period)
Description: The PASI 6-month AUC is a time adjusted total PASI score over the 6 month (180 days) period. The AUC is a continuous measurement (not a score on a scale); a lower value is considered better and a higher value is considered worse. The weighted average PASI score over 6 months (using all available PASI scores during a 6 month period [from Day 0 to 180 days]) is obtained by using PASI 6-month AUC /180 days.
Time Frame: Day 0 to 180 days
Population: Participants with at least two post Study P04563 randomization PASI scores (at least one is 150 days or more from Study P04563 randomization).
Measure: Mean (Standard Error); unit: 6-month PASI AUC
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Number analyzed (Participants) | 186 | 183
6-month PASI AUC | 566.2 (51.22) | 1098.0 (53.48)

5. Secondary Outcome: PASI 12-month AUC (Time Adjusted Total PASI Score Over the 12 Month Period)
Description: The PASI 12-month AUC is a time adjusted total PASI score over the 12 month (360 days) period. The AUC is a continuous measurement (not a score on a scale); and a lower value is considered better. The weighted average PASI score over 12 months (using all available PASI scores during a 12 month period [from Day 0 to 360 days]) is is obtained by using PASI 12-month AUC /360 days.
Time Frame: Day 0 to 360 days
Population: Participants with at least two post Study P04563 randomization PASI scores (at least one is 330 days or more from Study P04563 randomization).
Measure: Mean (Standard Error); unit: 12-month PASI AUC
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Number analyzed (Participants) | 105 | 91
12-month PASI AUC | 860.7 (92.46) | 2214.2 (108.5)

ADVERSE EVENTS:
Arm/Group | Maintenance Infliximab | Intermittent Infliximab
Serious Adverse Events (participants affected / at risk) | 24/222 | 23/219
Other Adverse Events (participants affected / at risk) | 95/222 | 97/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Infliximab (N=222) | Intermittent Infliximab (N=219)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
MACULAR HOLE (Eye disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 1 (1) | 8 (10)
POLYSEROSITIS (General disorders) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABSCESS JAW (Infections and infestations) | 1 (1) | 0 (0)
ACUTE TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
BIOPSY PROSTATE (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Infliximab (N=222) | Intermittent Infliximab (N=219)
INFUSION RELATED REACTION (General disorders) | 20 (43) | 25 (49)
NASOPHARYNGITIS (Infections and infestations) | 46 (67) | 48 (64)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22 (33) | 30 (40)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (15) | 11 (14)
HEADACHE (Nervous system disorders) | 14 (24) | 23 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's representative will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.